CLINICAL TRIAL: NCT00813371
Title: Airway Pressure Release Ventilation as a Preventative Strategy in Patients at Risk for Acute Respiratory Distress Syndrome
Brief Title: Airway Pressure Release Ventilation as a Preventative Strategy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left the institution before subjects were enrolled
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Jack Shannon, M.D., Texas Tech University Health Sciences Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TTUHSC-L08-152
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Lung Injury; Respiratory Failure; Trauma
Keywords: Acute Respiratory Distress Syndrome; acute lung injury; Airway Pressure Release Ventilation; ARDSnet; Bi-level; respiratory failure; trauma; APRV
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury; Respiratory Insufficiency; Wounds and Injuries | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Airway Pressure Release Ventilation Arm
  Interventions: Device: Airway Pressure Release Ventilation
- 2 (Active Comparator): ARDSnet protocol
  Interventions: Device: ARDSnet protocol

INTERVENTIONS:
Device: Airway Pressure Release Ventilation — Airway Pressure Release Ventilation (APRV) also known as Bi-Vent or Bi-Level ventilation is a time-cycled, pressure-limited mode of ventilation that allows spontaneous respiration throughout the ventilator cycle.
  Arms: 1
Device: ARDSnet protocol — ARDSnet protocol
  Arms: 2

SUMMARY:
The early initiation of Airway Pressure Release Ventilation in multi-system trauma patients decreases the incidence and severity of acute lung injury and Acute Respiratory Distress Syndrome and allows faster recovery of lung function.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients age 16 or older
* Trauma patients requiring ventilatory support within 48 hours of injury
* Those with anticipated ventilatory support ≥ 24 hours
* Subject or authorized representative (AR) has signed an informed consent form (ICF)
* Subjects age 16 or 17 who have signed an assent document and/or AR has signed an ICF

Exclusion Criteria:

* Significant chronic lung disease defined as lung pathology requiring home O2 use
* Chronic heart disease defined as NYHC III or higher
* Persistent bronchopulmonary air leak
* Contraindications to permissive hypercapnia (ex. Intracerebral bleeding, brain tumor, fulminant hepatic failure, and hemodynamic instability)
* Pulmonary artery occlusion pressures ≥ 18 mmHg
* Severe neurologic injury that may prevent the patient from having a reasonable opportunity for weaning as determined by the clinical study team
* Immuno-compromised patients secondary to drugs or disease
* Neuromuscular disease that impairs ability to ventilate spontaneously (ex. Spinal injury at or above C5, ALS, Guillain-Barre syndrome, Myasthenia Gravis)
* History of pneumonectomy
* Pregnancy
* Burns with TBSA ≥ 20%
* Acute MI as the cause of ALI/ARDS
* All other contraindications to APRV
* Patients who cannot be randomized within 12 hours of intubation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the number of ventilator-free days. | from randomization to study termination

SECONDARY OUTCOMES:
effects of ventilator mode on ventilation | duration of ventilatory assistance
duration of ICU stay | time in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Jack Shannon, M.D., Principal Investigator — Texas Tech University Health Sciences Center; John Griswold, M.D., Study Director — Texas Tech University Health Sciences Center